CLINICAL TRIAL: NCT00841555
Title: A Phase I Trial of Hypofraction Radiotherapy + Temozolomide in the Treatment of Patients With Glioblastoma Multiforme and Anaplastic Astrocytoma of the Brain
Brief Title: Temozolomide and Radiation Therapy in Treating Patients With Newly Diagnosed Glioblastoma Multiforme or Anaplastic Astrocytoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-08119; NCI-2011-03149 (Registry Identifier: Clinical Trial Reporting Program (CTRP))
Record Dates: First submitted 2009-02-10; First posted 2009-02-11 (Estimated); Results first posted 2016-04-27 (Estimated); Last update posted 2018-04-18 (Actual); Status verified 2018-04

CONDITIONS: Glioblastoma Multiforme/Anaplastic Astrocytoma
Keywords: adult giant cell glioblastoma; adult gliosarcoma; adult anaplastic astrocytoma; adult glioblastoma; GBM/AA
MeSH Terms: conditions — Glioblastoma; Astrocytoma; Gliosarcoma | interventions — Temozolomide; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Hypofractionation Radiotherapy+Temozolomide (Experimental): Patients will receive temozolomide PO daily for 5 weeks. Beginning week 1 after initiation of temozolomide therapy, patients undergo HIMRT times a week for a total of 15 fractions.
  Interventions: Drug: temozolomide; Radiation: Hypofractionated radiation therapy; Radiation: Intensity-modulated radiation therapy

INTERVENTIONS:
Drug: temozolomide — Chemotherapy will be given for 5 weeks; it will start 1 week before Radiotherapy, will continue for the 3 weeks of Radiotherapy, and will continue for 1 week post-Radiotherapy.
  Dose Level 1: 50 mg/m2 x first 4 weeks/75 mg/m2 x last 1 weeks of treatment Dose Level 2: 65 mg/m2 x first 4 weeks/75 mg/m2 x last 1 weeks of treatment Dose Level 3: 75 mg/m2 over the entire 5 weeks of treatment
  Other Names: Temodar; Temodal
Radiation: Hypofractionated radiation therapy — Patients will undergo HIMRT
Radiation: Intensity-modulated radiation therapy — Patients undergo HIMRT
  Other Names: IMRT

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as temozolomide, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Radiation therapy uses high-energy x-rays to kill tumor cells. Specialized radiation therapy that delivers a high dose of radiation directly to the tumor may kill more tumor cells and cause less damage to normal tissue. Giving chemotherapy together with radiation therapy may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of temozolomide when given together with radiation therapy in treating patients with newly diagnosed glioblastoma multiforme or anaplastic astrocytoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the maximum tolerated dose of temozolomide when given in combination with hypofractionated intensity-modulated conformal stereotactic radiotherapy in patients with newly diagnosed de novo glioblastoma multiforme or anaplastic astrocytoma.

Secondary

* To determine the time to neuroradiological evidence of tumor recurrence or progression in patients treated with this regimen.
* To determine the survival time of patients treated with this regimen.
* To determine the time spent in a Karnofsky performance status of 60-100%.

OUTLINE: This is a dose-escalation study of temozolomide.

Beginning 1-3 weeks following surgery or biopsy, patients receive oral temozolomide once daily for 5 weeks. Beginning 1 week after starting temozolomide, patients also undergo hypofractionated intensity-modulated conformal stereotactic radiotherapy once daily 5 days a week for 3 weeks.

After completion of study treatment, patients are followed at 1 month, 2 months, and 3 months, and then every 3 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have De novo glioblastoma multiforme, anaplastic astrocytoma, anaplastic oligodendrogliomas, mixed anaplastic oligoastrocytomas, gliosarcoma of the Brain, not involving the brain stem or optics chiasm, diagnosed following biopsy or tumor removal.
* Age > 18 years
* Given written consent
* Adequate bone marrow reserve(hemoglobin > 10 grams, Absolute neutrophil count > 1500 / mm3, platelets > 100,000/ mm3)
* Normal renal function(BUN < 24 mg/dL, Creatinine < 1.3 mg/dL)
* Normal liver function(Total Bilirubin < 1.5 mg/dL, SGPT/ALT < 60 U/L)

Exclusion Criteria:

* Have a Karnofsky score of < 60 [Appendix B] or age < 18 years.
* Prior chemotherapy and/or radiotherapy of their glioblastomamultiforme, anaplastic astrocytoma, anaplastic oligodendrogliomas, mixed anaplastic oligoastrocytomas, gliosarcoma.
* Tumors located in the brainstem or optic chiasm.
* Prior radiation therapy to the brain
* Prior chemotherapy within the past 6 weeks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2009-02-13 (Actual); Primary Completion 2013-02-13 (Actual); Study Completion 2014-11-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mario Ammirati, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

REFERENCES:
- [Result] Ammirati M, Chotai S, Newton H, Lamki T, Wei L, Grecula J. Hypofractionated intensity modulated radiotherapy with temozolomide in newly diagnosed glioblastoma multiforme. J Clin Neurosci. 2014 Apr;21(4):633-7. doi: 10.1016/j.jocn.2013.09.005. Epub 2013 Oct 3. PMID 24380758
- See also: Jamesline — http://cancer.osu.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled between 2009 and 2012
Groups:
- Dose Level 1: 50 mg/m2: Patients will receive temozolomide PO daily for 5 weeks. Beginning week 1 after initiation of temozolomide therapy, patients undergo HIMRT times a week for a total of 15 fractions.
  temozolomide: Chemotherapy will be given for 5 weeks; it will start 1 week before Radiotherapy, will continue for the 3 weeks of Radiotherapy, and will continue for 1 week post-Radiotherapy.
  Dose Level 1: 50 mg/m2 x first 4 weeks/75 mg/m2 x last 1 weeks of treatment
  Hypofractionated radiation therapy: Patients will undergo HIMRT
  Intensity-modulated radiation therapy: Patients undergo HIMRT
- Dose Level 2: 65 mg/m2: Patients will receive temozolomide PO daily for 5 weeks. Beginning week 1 after initiation of temozolomide therapy, patients undergo HIMRT times a week for a total of 15 fractions.
  temozolomide: Chemotherapy will be given for 5 weeks; it will start 1 week before Radiotherapy, will continue for the 3 weeks of Radiotherapy, and will continue for 1 week post-Radiotherapy.
  Dose Level 2: 65 mg/m2 x first 4 weeks/75 mg/m2 x last 1 weeks of treatment
  Hypofractionated radiation therapy: Patients will undergo HIMRT
  Intensity-modulated radiation therapy: Patients undergo HIMRT
- Dose Level 3: 75 mg/m2: Patients will receive temozolomide PO daily for 5 weeks. Beginning week 1 after initiation of temozolomide therapy, patients undergo HIMRT times a week for a total of 15 fractions.
  temozolomide: Chemotherapy will be given for 5 weeks; it will start 1 week before Radiotherapy, will continue for the 3 weeks of Radiotherapy, and will continue for 1 week post-Radiotherapy.
  Dose Level 3: 75 mg/m2 over the entire 5 weeks of treatment
  Hypofractionated radiation therapy: Patients will undergo HIMRT
  Intensity-modulated radiation therapy: Patients undergo HIMRT
Period: Overall Study
Arm/Group | Dose Level 1: 50 mg/m2 | Dose Level 2: 65 mg/m2 | Dose Level 3: 75 mg/m2
Started | 3 | 3 | 3
Completed | 3 | 3 | 3
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Glioblastoma multiforme (GBM) patients
Groups:
- Dose Level 1: Patients will receive temozolomide PO daily for 5 weeks. Beginning week 1 after initiation of temozolomide therapy, patients undergo HIMRT times a week for a total of 15 fractions.
  temozolomide: Chemotherapy will be given for 5 weeks; it will start 1 week before Radiotherapy, will continue for the 3 weeks of Radiotherapy, and will continue for 1 week post-Radiotherapy.
  Dose Level 1: 50 mg/m2 x first 4 weeks/75 mg/m2 x last 1 weeks of treatment
  Hypofractionated radiation therapy: Patients will undergo HIMRT
  Intensity-modulated radiation therapy: Patients undergo HIMRT
- Dose Level 2: Patients will receive temozolomide PO daily for 5 weeks. Beginning week 1 after initiation of temozolomide therapy, patients undergo HIMRT times a week for a total of 15 fractions.
  temozolomide: Chemotherapy will be given for 5 weeks; it will start 1 week before Radiotherapy, will continue for the 3 weeks of Radiotherapy, and will continue for 1 week post-Radiotherapy.
  Dose Level 2: 65 mg/m2 x first 4 weeks/75 mg/m2 x last 1 weeks of treatment
  Hypofractionated radiation therapy: Patients will undergo HIMRT
  Intensity-modulated radiation therapy: Patients undergo HIMRT
- Dose Level 3: Patients will receive temozolomide PO daily for 5 weeks. Beginning week 1 after initiation of temozolomide therapy, patients undergo HIMRT times a week for a total of 15 fractions.
  temozolomide: Chemotherapy will be given for 5 weeks; it will start 1 week before Radiotherapy, will continue for the 3 weeks of Radiotherapy, and will continue for 1 week post-Radiotherapy.
  Dose Level 3: 75 mg/m2 over the entire 5 weeks of treatment
  Hypofractionated radiation therapy: Patients will undergo HIMRT
  Intensity-modulated radiation therapy: Patients undergo HIMRT
- Total: Total of all reporting groups
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3 | Total
Number analyzed (Participants) | 3 | 3 | 3 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 0 | 2 | 4
  >=65 years | 1 | 3 | 1 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 0 | 3
  Male | 1 | 2 | 3 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 3 | 3 | 9
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 3 | 3 | 3 | 9
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: patients]
  United States | 3 | 3 | 3 | 9

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose(MTD)of Temozolomide(TMZ)
Description: This study is designed as a phase I dose escalation trial using the Standard Method of dose escalation of three patients per dose level to determine the MTD of TMZ (up to 75 mg/m 2 /day) when TMZ is used with HIMRT for patients with glioblastoma multiforme(GBM) or Anaplastic Astrocytoma(AA)of the brain. The 3 dose levels will be evaluated using the standard method to determine if either represents an MTD based on DLT. If DLT is not observed at all doses level, the greater of the three levels will be recommended for phase II evaluations of treatment effect.
Time Frame: up to 12-16 months
Measure: Number; unit: mg/m^2
Groups:
- Hypofractionation Radiotherapy+Temozolomide: Patients will receive temozolomide PO daily for 5 weeks. Beginning week 1 after initiation of temozolomide therapy, patients undergo HIMRT times a week for a total of 15 fractions.
  temozolomide: Chemotherapy will be given for 5 weeks; it will start 1 week before Radiotherapy, will continue for the 3 weeks of Radiotherapy, and will continue for 1 week post-Radiotherapy.
  Dose Level 1: 50 mg/m2 x first 4 weeks/75 mg/m2 x last 1 weeks of treatment Dose Level 2: 65 mg/m2 x first 4 weeks/75 mg/m2 x last 1 weeks of treatment Dose Level 3: 75 mg/m2 over the entire 5 weeks of treatment
  Hypofractionated radiation therapy: Patients will undergo HIMRT
  Intensity-modulated radiation therapy: Patients undergo HIMRT
Arm/Group | Hypofractionation Radiotherapy+Temozolomide
Number analyzed (Participants) | 9
mg/m^2 | 75

2. Secondary Outcome: Time to Neuroradiological Evidence of Tumor Recurrence or Progression
Description: As a small phase I study, no inferential statistical tests of hypotheses are planned. Data collected will be providing descriptive summary statistics. However, these estimates will allow statistically sound experimental designs and sample size calculations for subsequent studies of therapeutic effect.
Time Frame: up to 12-16 months
Reporting Status: Not Posted

3. Secondary Outcome: Survival Time
Description: All patients will be followed to death. Active follow-up with disease evaluation with scans will be terminated if the patient's physician deems it in the patient's interest not to continue or upon patient request.
Time Frame: up to 2 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Hypofractionation Radiotherapy+Temozolomide
Number analyzed (Participants) | 9
months | 12.7 [2.5 to 17.6]

4. Secondary Outcome: Time Spent in a Karnofsky Performance Status of 60-100%
Description: Time spent in a KPS ≥70 was calculated from the date of diagnosis of Karonofsky Performance Status decline (KPS<70) or censored at the last date the patient was known with KPS ≥70. The KPS higher scores indicates normal activity status.
Time Frame: up to 12-16 months
Population: Kaplan-Meier analysis for time spent in a Karnofsky performance status (KPS) ≥70
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Hypofractionation Radiotherapy+Temozolomide
Number analyzed (Participants) | 9
months | 8.1 [2.4 to 15.6]

ADVERSE EVENTS:
Description: The National Cancer Institute Common Terminology for Adverse Events (CTCAE) 3.0 was utilized for grading patients adverse events.
Groups:
- 50 mg/m2: Patients will receive temozolomide PO daily for 5 weeks. Beginning week 1 after initiation of temozolomide therapy, patients undergo HIMRT times a week for a total of 15 fractions.
  temozolomide: Chemotherapy will be given for 5 weeks; it will start 1 week before Radiotherapy, will continue for the 3 weeks of Radiotherapy, and will continue for 1 week post-Radiotherapy.
  Dose Level 1: 50 mg/m2 x first 4 weeks/75 mg/m2 x last 1 weeks of treatment
  Hypofractionated radiation therapy: Patients will undergo HIMRT
  Intensity-modulated radiation therapy: Patients undergo HIMRT
- 65 mg/m2: Patients will receive temozolomide PO daily for 5 weeks. Beginning week 1 after initiation of temozolomide therapy, patients undergo HIMRT times a week for a total of 15 fractions.
  temozolomide: Chemotherapy will be given for 5 weeks; it will start 1 week before Radiotherapy, will continue for the 3 weeks of Radiotherapy, and will continue for 1 week post-Radiotherapy.
  Dose Level 2: 65 mg/m2 x first 4 weeks/75 mg/m2 x last 1 weeks of treatment Hypofractionated radiation therapy: Patients will undergo HIMRT
  Intensity-modulated radiation therapy: Patients undergo HIMRT
- 75 mg/m2: Patients will receive temozolomide PO daily for 5 weeks. Beginning week 1 after initiation of temozolomide therapy, patients undergo HIMRT times a week for a total of 15 fractions.
  temozolomide: Chemotherapy will be given for 5 weeks; it will start 1 week before Radiotherapy, will continue for the 3 weeks of Radiotherapy, and will continue for 1 week post-Radiotherapy.
  Dose Level 3: 75 mg/m2 over the entire 5 weeks of treatment
  Hypofractionated radiation therapy: Patients will undergo HIMRT
  Intensity-modulated radiation therapy: Patients undergo HIMRT
Arm/Group | 50 mg/m2 | 65 mg/m2 | 75 mg/m2
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 3/3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 50 mg/m2 (N=3) | 65 mg/m2 (N=3) | 75 mg/m2 (N=3)
Fatigue (General disorders) | 3 (3) | 2 (2) | 2 (2)
Headache (Nervous system disorders) | 1 (1) | 2 (2) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 3 (3)
Partial seizure (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Motor deficits (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Numbness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Vision changes (Eye disorders) | 2 (2) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Memory deficits (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Confusion (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Stomach cramps (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
High ALT (Investigations) | 1 (1) | 1 (1) | 2 (2)
Low Calcium (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
High gluclose (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Thrombocytopenia (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes